CLINICAL TRIAL: NCT02818439
Title: Anticipating and Tracking: Pack of Gerontological Assessment Embedded
Acronym: ARPEGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PO12141*
Record Dates: First submitted 2016-06-16; First posted 2016-06-29 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Elderly
Keywords: Old person

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: evaluation of frailty

SUMMARY:
ARPEGE project fits within the general framework of maintaining functional autonomy in the frail elderly. The early identification of elderly people at risk of frailty is essential to be able to make corrective actions to maintain a quality of life desired by the person. ARPEGE offers tracking and monitoring based on a corpus mobile evaluation of frailty, that could be used in various environments (home, prevention center, office of the general practitioner, geriatric consultation), and manipulated intuitively by professionals not specialists.

This four-year project spearheaded by the University of technology of Troyes in partnership with the University of Reims Champagne-Ardenne also brings a set of partners and experts in the region and outside, so that the proposed solution has the qualities necessary for its deployment in terms of value diagnostic, use, acceptability and perfectly controlled ethics.

The Region has made "longevity aging" theme one of its priorities. This image of driver of innovation in this area can only be enhanced by a program like ARPEGE. Beyond the scientific and technological results expected, one can imagine the potential socio-economic benefits if this tracking solution is deployed on a large scale.

ELIGIBILITY:
Inclusion Criteria:

* 70 years or older
* GIR 4, 5 or 6
* Consenting to participate in the study

Exclusion Criteria:

* Severe cognitive impairment ( MMSE < 10)
* Major neurosensory disorders
* Full hospitalization or not (acute care and rehabilitation..)
* Non- affiliation to a social security scheme
* Major protected by law (guardianship, trusteeship)
* Informed consent not provide

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 216 (Actual)
Dates: Start 2013-10-14 (Actual); Primary Completion 2014-10-14 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Duke Health Profile: Quality of life questionnaire | up to 36 months
  The Duke Health Profile is a generic health-related quality of life questionnaire that comprises 17 items grouped in 10 scales: physical health, mental health, social health, general health (aggregate score of the 3 previous scales), perceived health, self-esteem, anxiety, depression, pain, and disability.
  Scores of each scale range from 0 to 100, with 100 representing optimum quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France